CLINICAL TRIAL: NCT02417935
Title: A Japan Post-Marketing, Randomized, Double-Blind, Parallel-Group, Flexible Dose Comparative Study to Assess the Non-Inferiority of Duloxetine Compared With Pregabalin in Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: A Study of Duloxetine (LY248686) in Participants With Diabetic Peripheral Neuropathic Pain (DPNP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14378; F1J-JE-HMHA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): 20 milligrams (mg) duloxetine orally once a day (QD) for one week and then 40 mg duloxetine orally QD for 3 weeks. Duloxetine dosage may be increased up to 60 mg QD at week 4 or week 8. Placebo will be given with duloxetine for blinding. Dosage will be tapered down during the final week of the study.
  Interventions: Drug: Duloxetine; Drug: Placebo
- Pregabalin (Active Comparator): 150 mg pregabalin orally twice a day (BID) for 1 week and then 300 mg pregabalin orally BID for 3 weeks. Pregabalin dosage may be increased up to 450 mg BID at week 4 or 8, and increased up to 600 mg BID at week 8. Placebo will be given with pregabalin for blinding. Dosage will be tapered down during the final week of the study.
  Interventions: Drug: Pregabalin; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: LY248686
  Arms: Duloxetine
Drug: Pregabalin — Administered orally
  Arms: Pregabalin
Drug: Placebo — Administered orally

SUMMARY:
The main purpose of this study is to evaluate the effectiveness and safety of the study drug known as duloxetine in participants with diabetic peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants present with pain due to bilateral, peripheral neuropathy
* Participants who have hemoglobin A1c (HbA1c) ≤9.4% (National Glycohemoglobin Standardization Program [NGSP]) at screening
* Participants who have HbA1c that has been measured 42 to 70 days prior to screening, and the range of variation in the values measured, thereafter, is within ±1.0% of the value measured at screening
* Participants who have a score of at least 4 on the mean of the 24-hour average pain score measured using 11-point NRS (Numeric Rating Scale) in the daily diary (should be calculated from records 7 days immediately prior to randomization)
* Participants who have made complete daily diary entries 80% or more of the time from screening to randomization

Exclusion Criteria:

* Participants who have undergone renal transplant, or are currently undergoing renal dialysis
* Participants who have uncontrolled narrow-angle glaucoma, history of uncontrolled seizures, or uncontrolled or poorly controlled hypertension
* Participants whose glycemic control has been poor within 70 days immediately prior to screening (for example, ketoacidosis requiring hospitalization, or hypoglycemia that may cause consciousness disorder)
* Pregnant or lactating female participants, or male participants who are planning for their partners to be or become pregnant during the timeframe of the study
* Participants who have hypersensitivity to multiple medications
* Participants who answered "yes" to either question 4 (active suicidal ideation with some intent to act, without specific plan) or question 5 (active suicidal ideation with specific plan and intent) on the "suicidal ideation" portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) or answered "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "suicidal behavior" portion of the C-SSRS; and the ideation or behavior occurred within the past month
* Participants who have past history of psychiatric diseases, such as depression, anxiety disorder, eating disorder, etc., that required drug therapy in the past 1 year, or who are currently having complications of these diseases or any history of manic psychosis or bipolar disorder
* Participants who have major depressive disorder as determined using the depression module of the Mini-International Neuropsychiatric Interview (MINI)
* Participants who have complications of diseases that are considered to affect the assessment of diabetic peripheral neuropathic pain. For example, nerve diseases with pain other than diabetic peripheral neuropathic pain (cervical spondylosis, carpal tunnel syndrome, spinal canal stenosis, and post-herpetic pain), pain diseases other than nerve diseases (collagen diseases, gout, chronic obstructive arteriosclerosis, and arthritis), and other pain at the site of evaluation (skin diseases and traumatic injury) are excluded
* Participants who have neuropathic pain suspected to be caused by alcohol
* Participants who have been treated with a monoamine oxidase (MAO) inhibitor(s) within 14 days immediately prior to randomization. Participants who visited the investigator site 14 days prior to randomization, those who have been treated with MAO inhibitors(s), thereafter, are excluded
* Participants who have alanine aminotransferase (ALT) and aspartate aminotransferase (AST) at a level ≥100 units/liter at screening
* Participants who have total bilirubin at a level ≥1.5 milligrams/deciliter (mg/dL) at screening
* Participants who have creatinine clearance (CrCL), calculated by Cockcroft-Gault, that is <1.0 milliliters/second (mL/s) (<60 mL/minute) at screening
* Participants who have a white blood cell (WBC) value <2500/cubic millimeters (mm3), neutrophils <1500/mm3, or platelets <100×103/mm3 on their hematology tests at screening
* Participants who are introduced to any treatments for diabetes, or a change in dosing regimen of any treatments for diabetes (exclude insulin treatment), or resumption of insulin treatment after screening
* Participants who have been treated with prohibited concomitant drug(s), or who have undergone prohibited concomitant treatment(s) after screening
* Participants who have taken restricted concomitant drugs 27 days immediately before screening, with continued use of the restricted concomitant drug prior to screening
* Participants who have taken acetaminophen for 4 days or more 7 days immediately prior to randomization

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05-13 (Actual); Study Completion 2017-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Enomoto H, Yasuda H, Nishiyori A, Fujikoshi S, Furukawa M, Ishida M, Takahashi M, Tsuji T, Yoshikawa A, Alev L. Duloxetine in patients with diabetic peripheral neuropathic pain in Japan: a randomized, doubleblind, noninferiority comparative study with pregabalin. J Pain Res. 2018 Sep 13;11:1857-1868. doi: 10.2147/JPR.S170646. eCollection 2018. PMID 30271191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 week Treatment period, followed by 1 week Tapering period, followed by 1 week follow-up period.
Groups:
- Pregabalin: Participants received flexible doses of 150 to 600 mg pregabalin orally twice a day (BID) along with Duloxetine placebo during treatment period.
  Participants who received higher doses of Pregabalin in treatment period received gradually the lower doses of Pregabalin along with Duloxetine placebo during tapering period.
- Duloxetine: Participants received flexible doses of 20 to 60 mg Duloxetine orally once a day (QD) along with Pregabalin placebo during treatment period.
  Participants who received higher doses of Duloxetine in treatment period received gradually the lower doses of Duloxetine along with Pregabalin placebo during tapering period.
Period: Treatment Period
Arm/Group | Pregabalin | Duloxetine
Started | 151 | 153
Received at Least One Dose of Study Drug | 151 | 152
Completed | 130 | 137
Not Completed | 21 | 16
Not completed — Adverse Event | 12 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Entry Criteria not met | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 3 | 1
Period: Tapering Period
Arm/Group | Pregabalin | Duloxetine
Started | 134 (Participants who discontinued treatment period had an option to enter the taper period) | 142 (Participants who discontinued treatment period had an option to enter the taper period)
Completed | 134 | 142
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Duloxetine | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.84) | 59.3 (8.16) | 59.6 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 109 | 111 | 220
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 151 | 152 | 303
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 151 | 152 | 303
Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — 24-hour average pain, night pain & 24-hour worst pain severity scores were recorded on an 11-point NRS, ranging from 0 (no pain) to 10 (pain as bad as you can imagine).Weekly mean was calculated based on daily score and used for the analysis.
  units on a scale
    Average Pain Score | 5.35 (1.129) | 5.38 (1.079) | 5.37 (1.102)
    Night Pain Score | 4.61 (1.855) | 4.92 (1.650) | 4.76 (1.759)
    Worst Pain Score | 6.25 (1.311) | 6.22 (1.237) | 6.23 (1.273)
Brief Pain Inventory - Short Form (BPI-SF) [Mean (Standard Deviation); unit: units on a scale] — BPI Severity (BPI-S) & BPI Interference Scores (BPI-I) are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (as bad as you can imagine) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
  units on a scale
    Worst Pain | 6.3 (1.45) | 6.3 (1.24) | 6.3 (1.35)
    Least Pain | 3.8 (1.74) | 3.9 (1.70) | 3.9 (1.72)
    Average Pain | 5.3 (1.21) | 5.3 (1.17) | 5.3 (1.19)
    Pain Right Now | 4.9 (1.60) | 4.9 (1.58) | 4.9 (1.59)
    General Activity | 3.1 (2.14) | 3.4 (2.21) | 3.3 (2.18)
    Mood | 3.3 (2.32) | 2.9 (2.23) | 3.1 (2.28)
    Walking Ability | 2.9 (2.28) | 2.8 (2.51) | 2.8 (2.39)
    Normal Work | 2.6 (2.11) | 2.6 (2.41) | 2.6 (2.26)
    Relations With Other People | 1.4 (1.81) | 1.4 (1.81) | 1.4 (1.80)
    Sleep | 2.7 (2.39) | 2.8 (2.37) | 2.8 (2.38)
    Enjoyment of Life | 2.6 (2.27) | 2.5 (2.24) | 2.5 (2.25)
    Average Interference Score | 2.66 (1.744) | 2.63 (1.875) | 2.64 (1.807)
Beck Depression Inventory-II (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory-II: BDI-II is a 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to symptoms of depression were scored on a 4-point scale ranging from 0 to 3 and was summed to give a single score. A total score of 0-13 was considered minimal range, 14-19 was mild, 20-28 was moderate, and 29-63 was severe.
  units on a scale | 6.2 (5.41) | 6.8 (5.90) | 6.5 (5.66)
Neuropathic Pain Symptom Inventory (NPSI) [Mean (Standard Deviation); unit: units on a scale] — NPSI questionnaire is a 12-item self-administered questionnaire that will be completed by the patient. It assesses 5 different dimensions of neuropathic pain: burning spontaneous pain, pressing spontaneous pain, paroxysmal pain, evoked pain, and paresthesias/dysesthesias. The NPSI includes 12 items: 10 descriptors of the different symptoms and 2 items for assessing the duration of spontaneous ongoing and paroxysmal pain. A total intensity score can be calculated as the sum of the scores of the 10 descriptors. (range: 0 (no pain) -100 (worst imaginable pain)).
  units on a scale | 31.8 (15.60) | 32.1 (16.49) | 31.9 (16.03)
EuroQol 5 Dimension (EQ-5D) [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D is a self-reported, 5-item scale used to assess the patient's health utility (mobility, self-care, usual activities, pain and discomfort, and depression/anxiety). Scoring is on a 3-point scale.These combinations of attributes were converted into a weighted health-state Index Score according to the Japan population-based algorithm.Range of the Index score is -0.111 - 1(higher score indicates better health state).
  units on a scale | 0.7253 (0.0903) | 0.7337 (0.1230) | 0.7296 (0.1079)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Weeks in the Weekly Mean of the 24-Hour Average Pain Score on the 11-Point Numeric Rating Scale (NRS)
Description: 11-point NRS measures the severity of pain over the previous 24 hours. Participants were asked to provide 24-hour average pain scores in the daily Participant diary and among these, the weekly mean of the 24-hour average pain score was calculated. Scores range from 0 (no pain) to 10 (pain as bad as you can imagine).
  Mixed Model Repeated Measures (MMRM) model with baseline value, Duration of diabetic peripheral neuropathic pain (DPNP), treatment, week, treatment-by-week interaction as fixed effects was used to produce Least Square Mean (LS Mean).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline observation for NRS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Pregabalin: Participants received flexible doses of 150 to 600 mg Pregabalin orally twice a day (BID) along with Duloxetine Placebo.
- Duloxetine: Participants received flexible doses of 20 to 60 mg Duloxetine orally once a day (QD) along with Pregabalin placebo.
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
units on a scale | -2.358 (0.133) | -2.286 (0.133)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Non-Inferiority — If the upper bound of the 95% CI does not exceed 0.51 (pre-defined non-inferiority margin), it will be concluded that duloxetine is not inferior to Pregabalin; p = 0.700, Mixed Models Analysis; Mean Difference (Final Values) = 0.072, 95% CI 2-sided [-0.295 to 0.439]

2. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at 12 Weeks
Description: PGI-I assessments was completed by the participant. The participant records how he/she perceives the degree of improvement (or worsening) at the time of assessment since taking treatment. The score ranges from 1 (very much better) to 7 (very much worse).
  MMRM model with duration of DPNP, treatment, visit, treatment-by-visit interaction as fixed effects was used to produce LS Mean.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had at least one post baseline observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
units on a scale | 2.6 (0.1) | 2.4 (0.1)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = 0.149, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

3. Secondary Outcome: Change From Baseline to 12 Weeks on the Brief Pain Inventory-Severity and Interference Rating Short Form (BPI-SF)
Description: Brief Pain Inventory Severity and Interference Scores: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (pain as bad as you can imagine) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
  MMRM model with baseline, duration of DPNP, treatment, visit, treatment-by-visit interaction as fixed effects was used to produce LS mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline observation for BPI-SF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
units on a scale
  Worst Pain | -2.8 (0.2) | -2.7 (0.2)
  Least Pain | -1.7 (0.1) | -1.9 (0.1)
  Average Pain | -2.5 (0.1) | -2.4 (0.1)
  Pain Right Now | -2.4 (0.1) | -2.4 (0.1)
  General Activity: number analyzed (Participants) | 149 | 151
  General Activity | -1.9 (0.1) | -2.1 (0.1)
  Mood: number analyzed (Participants) | 149 | 151
  Mood | -1.9 (0.1) | -2.1 (0.1)
  Walking Ability: number analyzed (Participants) | 149 | 151
  Walking Ability | -1.8 (0.1) | -1.9 (0.1)
  Normal Work: number analyzed (Participants) | 149 | 151
  Normal Work | -1.6 (0.1) | -1.8 (0.1)
  Relations with Other People: number analyzed (Participants) | 149 | 151
  Relations with Other People | -0.7 (0.1) | -0.9 (0.1)
  Sleep: number analyzed (Participants) | 149 | 151
  Sleep | -1.7 (0.1) | -1.7 (0.1)
  Enjoyment of Life: number analyzed (Participants) | 149 | 151
  Enjoyment of Life | -1.6 (0.1) | -1.8 (0.1)
  Average Interference | -1.60 (0.10) | -1.77 (0.10)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Worst Pain; Test type: Other; p = .535, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Least Pain; Test type: Other; p = .436, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 3: Comparison: Pregabalin vs Duloxetine; Average Pain; Test type: Other; p = .534, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.5]
Statistical Analysis 4: Comparison: Pregabalin vs Duloxetine; Pain Right Now; Test type: Other; p = .948, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; General Activity; Test type: Other; p = .225, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.1]
Statistical Analysis 6: Comparison: Pregabalin vs Duloxetine; Mood; Test type: Other; p = .276, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 7: Comparison: Pregabalin vs Duloxetine; Walking Ability; Test type: Other; p = .507, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Normal Work; Test type: Other; p = .216, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 9: Comparison: Pregabalin vs Duloxetine; Relations with other people; Test type: Other; p = .233, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 10: Comparison: Pregabalin vs Duloxetine; Sleep; Test type: Other; p = .857, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Enjoyment of life; Test type: Other; p = .133, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 12: Comparison: Pregabalin vs Duloxetine; Average Interference Score; Test type: Other; p = .246, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.44 to 0.11]

4. Secondary Outcome: Change From Baseline to 12 Weeks on the Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI questionnaire is a 12-item self-administered questionnaire that will be completed by the participant. It assesses 5 different dimensions of neuropathic pain on a scale of 0 (no symptom) to 10 (worst imaginable symptom): burning spontaneous pain, pressing spontaneous pain, paroxysmal pain, evoked pain, and paresthesias/dysesthesias. The NPSI includes 12 items: 10 descriptors of the different symptoms and 2 items for assessing the duration of spontaneous ongoing and paroxysmal pain. A total score can be calculated as the sum of the scores of the 10 descriptors with scale range: 0 (no pain) -100 (worst pain imaginable).
  Analysis of Covariance (ANCOVA) model with last observation carried forward (LOCF) with baseline, treatment, and duration of DPNP as fixed effects was used to produce LS mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post-baseline observation for NPSI.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 148 | 151
units on a scale
  Total Score | -15.4 (1.1) | -16.1 (1.1)
  Burning Pain | -1.1 (0.2) | -1.3 (0.2)
  Pressing Pain | -1.4 (0.1) | -1.4 (0.1)
  Paroxysmal Pain | -1.7 (0.1) | -1.7 (0.1)
  Evoked Pain | -1.0 (0.1) | -1.2 (0.1)
  Paresthesia/Dysesthesia | -2.5 (0.1) | -2.6 (0.1)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Total Score; Test type: Other; p = .627, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.6 to 2.2]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Burning Pain; Test type: Other; p = .355, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 3: Comparison: Pregabalin vs Duloxetine; Pressing Pain; Test type: Other; p = .731, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 4: Comparison: Pregabalin vs Duloxetine; Paroxysmal Pain; Test type: Other; p = .721, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Evoked Pain; Test type: Other; p = .345, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 6: Comparison: Pregabalin vs Duloxetine; Paresthesia/Dysesthesia; Test type: Other; p = .557, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.3]

5. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at 12 Weeks
Description: CGI-I measures clinician's perception of participant improvement at the time of assessment (compared with the start of treatment) with scores ranging from 1 (very much better) to 7 (very much worse).
  MMRM model with duration of DPNP, treatment, visit and treatment-by-visit interaction as fixed effects was used to produce LS Mean.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had at least one post baseline observation for CGI-I
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
units on a scale | 2.6 (0.1) | 2.5 (0.1)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = .106, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0]

6. Secondary Outcome: Change From Baseline to 12 Weeks on the EuroQol 5 Dimension (EQ-5D)
Description: The EQ-5D is a self-reported, 5-item scale used to assess the patient's health utility (mobility, self-care, usual activities, pain and discomfort, and depression/anxiety). Scoring is on a 3-point scale.These combinations of attributes were converted into a weighted health-state Index Score according to the Japan population-based algorithm (range of the Index score is -0.111 - 1).A higher score indicates better health state.
  ANCOVA model with LOCF with baseline value, treatment and duration of DPNP as fixed effects was used to produce LS mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline observation for EQ-5D.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 148 | 151
units on a scale | 0.1004 (0.0112) | 0.1144 (0.0112)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = .361, ANCOVA; Mean Difference (Final Values) = 0.0140, 95% CI 2-sided [-0.0161 to 0.0441]

7. Secondary Outcome: Change From Baseline to 12 Weeks on the Beck Depression Inventory-II (BDI-II) Total Score
Description: Beck Depression Inventory-II: BDI-II is a 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to symptoms of depression were scored on a 4-point scale ranging from 0 to 3 and was summed to give a single score. A total score of 0-13 was considered minimal range, 14-19 was mild, 20-28 was moderate, and 29-63 was severe.
  MMRM model with baseline value, duration of DPNP, treatment, visit and treatment-by-visit interaction as fixed effects was used to produce LS mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline observation for BDI-II.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 146 | 141
units on a scale | -2.5 (0.3) | -2.3 (0.3)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = .701, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.1]

8. Secondary Outcome: Change From Baseline to 12 Weeks in the Weekly Mean of Night Pain Scores on the 11-Point NRS
Description: Night pain severity scores were recorded on an 11-point NRS in the daily patient diary, ranging from 0 (no pain) to 10 (pain as bad as you can imagine).The weekly mean of the night pain score was calculated based on the daily pain score.
  MMRM model with baseline value, treatment, week, duration of DPNP and treatment-by-week interaction as fixed effects was used to produce LS mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline observation for night pain NRS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
units on a scale | -2.166 (0.131) | -2.160 (0.131)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = .976, Mixed Models Analysis; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.355 to 0.366]

9. Secondary Outcome: Change From Baseline to 12 Weeks in the Weekly Mean of the 24-Hour Worst Pain Scores on the 11-Point NRS
Description: 24-hour worst pain severity scores were recorded on an 11-point NRS in the daily patient diary, ranging from 0 (no pain) to 10 (pain as bad as you can imagine).The weekly mean of the worst pain score was calculated based on the daily score.
  MMRM model with baseline value, duration of DPNP, treatment, week, treatment-by-week interaction as fixed effects was used to produce LS mean.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline observation for worst pain score NRS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
units on a scale | -2.553 (0.145) | -2.416 (0.145)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = .503, Mixed Models Analysis; Mean Difference (Final Values) = 0.136, 95% CI 2-sided [-0.264 to 0.537]

10. Secondary Outcome: Number of Participants With a 30% and 50% Reduction in the Weekly Mean of the 24-Hour Average Pain Score on the 11-Point NRS at 12 Weeks
Description: 11-point NRS measures the severity of pain over the previous 24 hours. Patients were asked to provide 24-hour average pain scores in the daily patient diary. scores range from 0 (no pain) to 10 (pain as bad as you can imagine) and among these, the weekly mean of the 24-hour average pain score was calculated based on daily score.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug & had baseline & at least one post-baseline observation for average pain score NRS .
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 149 | 152
Participants
  30% Reduction | 94 | 100
  50% Reduction | 62 | 62
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Test type: Other; p = .632, Fisher Exact — 30% reduction
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; 50% Reduction; Test type: Other; p = .907, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Arm/Group | Pregabalin | Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/152
Serious Adverse Events (participants affected / at risk) | 6/151 | 1/152
Other Adverse Events (participants affected / at risk) | 91/151 | 86/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=151) | Duloxetine (N=152)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=151) | Duloxetine (N=152)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6)
Diabetic gastroenteropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 12 (13)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (9)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Feeling abnormal (General disorders) | 4 (4) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2)
Nodule (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (3) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Myringitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (5)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 12 (13) | 9 (10)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 22 (22) | 9 (11)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 22 (23) | 19 (21)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (6):
  • Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT02417935/SAP_000.pdf
  • Study Protocol: Protocol (2014-05-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02417935/Prot_001.pdf
  • Study Protocol: Protocol Amendment (a) (2014-09-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT02417935/Prot_002.pdf
  • Study Protocol: Protocol Amendment (b) (2015-04-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT02417935/Prot_003.pdf
  • Study Protocol: Protocol Amendment (c) (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02417935/Prot_004.pdf
  • Study Protocol: Protocol Amendment (d) (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT02417935/Prot_005.pdf